CLINICAL TRIAL: NCT05035940
Title: FAA National Sleep Study on the Effects of Aircraft Noise on Sleep
Brief Title: Federal Aviation Administration (FAA) National Sleep Study
Acronym: NSS
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Federal Aviation Administration Office of Environment and Energy (Unknown); Harris Miller Miller & Hanson Inc. (Unknown); Westat (Other)
Responsible Party: Principal Investigator, Mathias Basner, MD, PhD, Professor, University of Pennsylvania
Other Study IDs: 833863
Record Dates: First submitted 2021-08-23; First posted 2021-09-05 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Noise Exposure
Keywords: Aircraft noise; Sleep disturbance
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This observational study will examine the relationship between aircraft noise exposure in the bedroom and objectively assessed sleep disturbance. Surveys will be mailed to randomly selected households around selected airports to recruit individuals for a 5 night in-home sleep study. Eligible survey respondents interested in participating in the sleep study will record nighttime indoor sounds using a portable audio recorder and wear a small device that collects heart rate and movement data for 5 consecutive nights. They will also complete brief morning questionnaires about their previous night's sleep and their sleep quality and a participant characteristics questionnaire. Collected data will be used to create an exposure-response model between aircraft noise exposure and sleep disturbance.

DETAILED DESCRIPTION:
Individuals who complete the recruitment survey, indicate their interest in participating in the study, and meet the eligibility criteria, will be enrolled in the 5-night in-home sleep study to collect noise and physiological (heart rate, body movements) measurements, and answer questionnaires about experiences during the previous night and a characteristics questionnaire that collects additional information relevant for sleep. After confirmation of eligibility and informed consent, subjects will be sent equipment by mail to measure body movements and ECG signals as well as sounds in the bedroom. Awakenings will be inferred from ECG and movement data using a previously validated algorithm, and analyzed relative to measured noise levels in the bedroom. The study nights will take place during the week, Monday night/Tuesday morning through Friday night/Saturday morning. Upon completion of the 5 nights, the questionnaires and equipment will be returned to the study team by mail. Survey mailing distribution, subject recruitment, and data collection for the in-home sleep study is expected to last 2 years, but may last up to 3 years.

The study population is adult residents of U.S. households who are exposed to relevant levels of nighttime air traffic (both in terms of number and sound pressure level of events) in communities in proximity to 77 airports that met the eligibility criteria for this study. Only areas with expected aircraft noise exposure levels of ≥40 decibels (dB) Lnight (average aircraft noise level during the nighttime period) outside were considered for the sample frame. To maximize the likelihood that there will be a range of indoor noise levels in the sample frame, the investigators will use probability sampling stratified on outdoor aircraft noise contour levels. For each of the selected 77 airports, noise exposure contour strata, were determined using the FAA's Aviation Environmental Design Tool and 2018 traffic data. These noise contours are based on Lnight and include the 40, 45, 50, and 55 dB contour to allow for stratified sampling from the following areas: 40<45, 45<50, 50<55, ≥55 dB. From each noise stratum, 100 subjects will be recruited into the in-home field study. Mailing addresses for the recruitment survey will be selected randomly from all households across the 77 airports within each of the 4 noise strata.

The primary study outcome is aircraft noise-induced awakening probability depending on the maximum sound pressure level of single aircraft events. Analyses will be weighted to better reflect the sampling universe, but unweighted analyses will also be performed. Secondary outcomes include, but are not limited to, self-reported sleep disturbance depending on noise metrics referring to longer time periods (i.e., last night or past year).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must currently live in a residence exposed to relevant levels of nocturnal aircraft traffic and have received a recruitment survey in the mail.
* Only one subject per household will be eligible, selected pseudo-randomly as the person in the household who most recently celebrated a birthday.
* In order to be eligible to participate in the in-home study, participants must have completed and returned the recruitment postal survey that was sent to their residence.

Exclusion Criteria:

Survey respondents interested in participating in the in-home sleep study are ineligible to participate if they:

* are less than 21 years of age;
* have a Body Mass Index (BMI) greater than 35 kg/m2 or less than 17 kg/m2;
* have been diagnosed with a sleep disorder, including obstructive or central sleep apnea, narcolepsy, restless legs syndrome, or periodic limb movement syndrome;
* frequently (3 or more times per week) use prescription or over the counter medication to aid sleep;
* have a hearing impairment;
* have a cardiac arrhythmia;
* work night shifts (defined as working for at least 4 hours between 00:00 to 06:00);
* have dependents that frequently require care during the night;
* are pregnant;
* previously participated in one of the pilot studies performed at Philadelphia airport or Atlanta airport; or
* habitually use earplugs or play back sounds in the bedroom that could mask aircraft noise.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is adult residents of U.S. households who are exposed to relevant levels of nighttime air traffic (both in terms of number and sound pressure level of events) in communities in proximity to an airport meeting the eligibility criteria for this study.
Sampling Method: Probability Sample
Enrollment: 401 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Noise-induced awakening | First 45 seconds of each aircraft noise event
  The probability of awakening (assessed with heart rate and body movements) depending on the maximum sound pressure level of an aircraft overflight (LAS,max measured inside the bedroom) during an aircraft noise event.

SECONDARY OUTCOMES:
Percent highly sleep disturbed | 1 year
  The recruitment survey contains a question: "Thinking about the last year or so, when you are here at home, how much does noise from aircraft disturb your sleep?" Subjects choosing "very" or "extremely" on the 5-point answer scale will be considered highly sleep disturbed. The investigators will investigate how long-term aircraft noise exposure metrics are associated with being highly sleep disturbed.

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Basner, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Perelman School of Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
Together with the sponsor, the study team is in the process of defining which data will be made available to the public after the end of the study in accordance with the Federal Records Retention Schedule.

REFERENCES:
- [Background] Smith MG, Rocha S, Witte M, Basner M. On the feasibility of measuring physiologic and self-reported sleep disturbance by aircraft noise on a national scale: A pilot study around Atlanta airport. Sci Total Environ. 2020 May 20;718:137368. doi: 10.1016/j.scitotenv.2020.137368. Epub 2020 Feb 17. PMID 32092522
- [Background] Smith MG, Witte M, Rocha S, Basner M. Effectiveness of incentives and follow-up on increasing survey response rates and participation in field studies. BMC Med Res Methodol. 2019 Dec 5;19(1):230. doi: 10.1186/s12874-019-0868-8. PMID 31805869
- [Background] Basner M, Witte M, McGuire S. Aircraft Noise Effects on Sleep-Results of a Pilot Study Near Philadelphia International Airport. Int J Environ Res Public Health. 2019 Aug 31;16(17):3178. doi: 10.3390/ijerph16173178. PMID 31480420